CLINICAL TRIAL: NCT04647201
Title: Study of Biomarkers in Blood and Tissue Samples of Septic Patients Complicated With Gastrointestinal Dysfunction
Brief Title: Study of Biomarkers in Patients of Sepsis Complicated With Gastrointestinal Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jianbo Yu (Other)
Responsible Party: Sponsor-Investigator, Jianbo Yu, Department of Anesthesiology, Director, Chief physician, Professor, Doctoral tutor, Tianjin Nankai Hospital
Organization: Tianjin Nankai Hospital (Other)
Other Study IDs: SGI-2020-11
Record Dates: First submitted 2020-11-22; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Sepsis; Gastrointestinal Dysfunction
Keywords: sepsis; gastrointestinal dysfunction; biomarkers
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Non-sepsis and non-GI adults
- Sepsis patients without GI: Patients who meet the criteria of sepsis3.0 with AGI grade I or less
- Sepsis patients with GI: Patients who meet the criteria of sepsis3.0 with AGI grade II or above

SUMMARY:
1. Title: Study of Biomarkers in Patients of Sepsis Complicated With Gastrointestinal Dysfunction
2. Research center: Single-center study.
3. Design of the research: A prospective and cohort study.
4. Object of the research: Patients with age≥18 years those who meet the diagnostic criteria of sepsis 3.0 complicated with GI and grouped into GI group and non-GI adults as control.
5. Sample size of the research: Not less than 30 patients in each group.
6. Research approach: After admission to ICU, patients were assigned to the indicated groups according to the criteria. In addition, blood samples were collected within 24 hours for detecting serum levels of HO-1, PINK1, PLK1as well as oxidative stress and inflammatory markers.For those who requiring intestinal surgery as treatment, the intestinal tissue specimens are retained.
7. Aim of the research: The find out the potential biomarkers in serum to help the diagnose and management of gastrointestinal dysfunction in septic patients.
8. Statistical analysis: Analytical study.
9. The estimated duration of the study#1-2 years.

DETAILED DESCRIPTION:
This study is a single-center, prospective, cohort study. In this study, the serum samples of septic patients complicated with or without GI are detected. The serum levels of HO-1, PINK1, PLK1as well as oxidative stress and inflammatory markers are compared in different groups. For those who requiring intestinal surgery as treatment, the intestinal tissue specimens are retained. Meanwhile, the clinical symptoms, intestinal motility indicators and intestinal barrier indicators are recorded. In addition, a biomarker model was established to provide important reference for diagnose and management of gastrointestinal dysfunction in septic patients.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Patients with sepsis who meet the criteria for sepsis 3.0
3. Patients complicated gastrointestinal dysfunction with AGI grade II or above
4. Agree to participate in this study and sign informed consent

Exclusion Criteria:

1. Refuse to participate in this study
2. Those who have chronic gastrointestinal diseases such as Crohn's disease and ulcerative colitis
3. Those who have recently used gastrointestinal motility drugs and within 5 times the half-life
4. Those who are participating in other drug clinical trials
5. Patient with HIV infection, patients in pregnancy or breast stage
6. In the opinion of the attending physician or researcher, there are other conditions that are not appropriate for the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with sepsis complicated with GI
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-11-23 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Multivariate data analysis of the metabolites | an average of one year
  Record the different metabolites between the control group and septic patients
Multivariate data analysis of the metabolites | an average of one year
  Record the different metabolites between the septic patient with or without GI

SECONDARY OUTCOMES:
Screening of differentially expressed metabolites as potential mortality predictors for sepsis complicated with GI | an average of one year
  Investigated the metabolites to distinguish the non-survivors from the survivors of sepsis complicated with GI

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Yu, PhD, Study Chair — Tianjin Nankai Hospital
Locations (1):
- Tianjin Nankai Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No
All of the individual participant data collected during the trial,after de-identification will be shared.And anyone who wishes to acess the date will beavailable for any purpose

REFERENCES:
- [Background] Assimakopoulos SF, Triantos C, Thomopoulos K, Fligou F, Maroulis I, Marangos M, Gogos CA. Gut-origin sepsis in the critically ill patient: pathophysiology and treatment. Infection. 2018 Dec;46(6):751-760. doi: 10.1007/s15010-018-1178-5. Epub 2018 Jul 12. PMID 30003491
- [Background] Reintam Blaser A, Poeze M, Malbrain ML, Bjorck M, Oudemans-van Straaten HM, Starkopf J; Gastro-Intestinal Failure Trial Group. Gastrointestinal symptoms during the first week of intensive care are associated with poor outcome: a prospective multicentre study. Intensive Care Med. 2013 May;39(5):899-909. doi: 10.1007/s00134-013-2831-1. Epub 2013 Jan 31. PMID 23370829
- [Background] Blaser A, Padar M, Tang J, Dutton J, Forbes A. Citrulline and intestinal fatty acid-binding protein as biomarkers for gastrointestinal dysfunction in the critically ill. Anaesthesiol Intensive Ther. 2019;51(3):230-239. doi: 10.5114/ait.2019.86049. PMID 31418255
- [Background] Reintam Blaser A, Regli A, De Keulenaer B, Kimball EJ, Starkopf L, Davis WA, Greiffenstein P, Starkopf J; Incidence, Risk Factors, and Outcomes of Intra-Abdominal (IROI) Study Investigators. Incidence, Risk Factors, and Outcomes of Intra-Abdominal Hypertension in Critically Ill Patients-A Prospective Multicenter Study (IROI Study). Crit Care Med. 2019 Apr;47(4):535-542. doi: 10.1097/CCM.0000000000003623. PMID 30608280
- [Background] Greis C, Rasuly Z, Janosi RA, Kordelas L, Beelen DW, Liebregts T. Intestinal T lymphocyte homing is associated with gastric emptying and epithelial barrier function in critically ill: a prospective observational study. Crit Care. 2017 Mar 22;21(1):70. doi: 10.1186/s13054-017-1654-9. PMID 28327177